CLINICAL TRIAL: NCT03909789
Title: Acute and Sustained Effects of Plant- Based Bio-Equivalent Nitrate Supplement Tablets on Blood Pressure Reduction, Nitric Oxide Mediated Endothelial Function and Saliva Bioconversion of Dietary Nitrate in Hypertensive Men and Women
Brief Title: Effect of Inorganic Nitrate Supplement on Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Matthew J. Budoff, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21835-01
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Blood Pressure; Endothelial Dysfunction
Keywords: Endothelium

STUDY DESIGN:
Intervention Model Description: Double Blind Placebo Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- plant based bioequivalent dietary nitrate supplement (Active Comparator): The nitrate supplement consists of nitrate-rich beetroot extract 20mg, thiamine mononitrate 90mg, potassium nitrate 480mg, ascorbic acid 150mg, folic acid 200mcg, methylcobalamin 200mcg, calcium 115mg, pomegranate fruit extract 5mg and green coffee bean extract 115mg.
  Interventions: Dietary Supplement: Plant based bioequivalent Nitrate supplementation
- placebo (Placebo Comparator): The Placebo does not contain any nitric oxide supplement.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Plant based bioequivalent Nitrate supplementation — The nitrate supplement consists of nitrate-rich beetroot extract 20mg, thiamine mononitrate 90mg, potassium nitrate 480mg, ascorbic acid 150mg, folic acid 200mcg, methylcobalamin 200mcg, calcium 115mg, pomegranate fruit extract 5mg and green coffee bean extract 115mg.
  Arms: plant based bioequivalent dietary nitrate supplement
Dietary Supplement: Placebo — Placebo
  Arms: placebo

SUMMARY:
The primary purpose of this project is to assess the efficacy (effectiveness) of plant-based nitrate tablets to elevate nitric oxide in your system as measured by saliva and effect on lowering blood pressure (BP), supporting blood vessel function in men and women with hypertension.

DETAILED DESCRIPTION:
This clinical trial is to assess the efficacy of plant-based bioequivalent Nitric Oxide supplement for improving blood pressure and endothelial reactivity over a 12 weeks intervention period in individuals with metabolic syndrome. The study also examines the effect of plant-based bioequivalent Nitric Oxide supplement on other markers of cardiovascular function and cardiovascular disease risk including Total, LDL and HDL-Cholesterol, Triglycerides, and a multitude of inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* age 40-75 years
* Hypertension >130/85 mmHg; men and women, 1:1 and stable medicated hypertensives
* Subjects must provide written informed consent after the scope and nature of the investigation has been explained to them

Exclusion Criteria:

* Any unstable medical, psychiatric or substance abuse disorder that in the opinion of the investigator or principal investigator is likely to affect the subject's ability to complete the study or precludes the subject's participation in the study
* Weight in excess of 250 pounds
* Bleeding disorder
* History of known coronary artery disease, myocardial infarction, stroke or life-threatening arrhythmia within the prior six months
* NYHA Class II- IV heart failure
* History of malignancy within the last 5 years (other than skin cancer) or evidence of active cancer which would require concomitant cancer chemotherapy
* Serum creatinine > 1.4 mg/dl
* Triglycerides > 400 at visit 1
* Drug or alcohol abuse, or current intake of more than 14 standard drinks per week
* Concurrent enrollment in another placebo-controlled trial
* Partial ileal bypass or known gastrointestinal disease limiting drug absorption
* Current tobacco use
* Current use of anticoagulants (except for anti-platelet agents)
* Renal failure
* History of hypertensive encephalopathy or cerebrovascular accident
* Hematological or biochemical values at screening outside the reference ranges considered as clinically significant in the opinion of the investigator or PI
* Pregnancy

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

PRIMARY OUTCOMES:
Rate of change in blood pressure | 12 weeks
  change in blood pressure (in millimeters of mercury) over twelve weeks under effect of active treatment and placebo

SECONDARY OUTCOMES:
changes in serum, plasma and salivary Nitrite and Nitrate | 12 weeks
  change in serum nitrate and nitrate levels (in mcg) over 12 weeks comparing active treatment to placebo
cardiometabolic relevant biomarkers (as compared to placebo) | 12 weeks
  measures of serum markers of inflammation (Crp) and glucose over 12 weeks in active vs placebo arms

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles Biomedical Research Institute at Harbor UCLA Medical Center, Torrance, California, United States

REFERENCES:
- [Derived] Cherukuri L, Birudaraju D, Kinninger A, Chaganti BT, Shekar C, Hamal S, Shaikh K, Flores F, Roy SK, Sotka W, Green SJ, Budoff MJ. Effect of a plant-based bioequivalent inorganic nitrate (NO3-) complex with vitamins, antioxidants and phytophenol rich food extracts in hypertensive individuals - A randomized, double-blind, placebo-controlled study. Clin Nutr ESPEN. 2020 Dec;40:327-335. doi: 10.1016/j.clnesp.2020.08.007. Epub 2020 Sep 7. PMID 33183558